CLINICAL TRIAL: NCT00146315
Title: Effectiveness of the Supervised Exercise for Patients With Coronary Heart Disease in the Primary Care Setting (ESCAP): a Randomized Clinical Trial
Brief Title: ESCAP: Supervised Exercise for Patients With Coronary Heart Disease in the Primary Care Setting
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Basque Health Service (Other Government)
Collaborators: Preventive Services and Health Promotion Research Network (Other); Castilla-La Mancha Health Service (Other); Castilla-León Health Service (Other); Dalt Sant Joan primary care center (Balears Islans Health Service) (Unknown); Public Health Service of Cataluña (Other); Public Health Service of Madrid (Other); Public Health Service of Galicia (Other); Cantabria Health Service (Other)
Responsible Party: Ricardo Ortega, Castilla La Mancha Health Service
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ESCAP-G03/170-200311075
Record Dates: First submitted 2005-09-06; First posted 2005-09-07 (Estimated); Last update posted 2011-06-01 (Estimated); Status verified 2011-05

CONDITIONS: Coronary Heart Disease
Keywords: Primary Health Care; Family Practice; Family Physician; Exercise; Coronary Heart Disease; Randomized Controlled Trials; Multicenter Studies
MeSH Terms: conditions — Coronary Disease; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (Active Comparator): Secondary prevention program for coronary heart disease
  Interventions: Behavioral: Secondary prevention program for coronary heart disease
- Supervised exercise (Experimental)
  Interventions: Behavioral: Supervised exercise on a stationary bicycle, 3-5 days a week

INTERVENTIONS:
Behavioral: Supervised exercise on a stationary bicycle, 3-5 days a week — Supervised exercise on a stationary bicycle, 3-5 days a week, plus a secondary prevention program for coronary heart disease
  Arms: Supervised exercise
Behavioral: Secondary prevention program for coronary heart disease — Secondary prevention program for coronary heart disease
  Arms: Control

SUMMARY:
In Spain, family physician are currently recommended to prescribe an unsupervised walking program to their coronary heart disease (CHD) patients as a part of their cardiac rehabilitation program. However, there are a few family physicians who provide their CHD patients with supervised exercise (30 minutes of pedaling on an stationary bicycle at 60-85% of the peak heart rate (HR) attained at the maximal or symptom limited treadmill test, 3 times a week) at their primary care health centers, thinking that these patients improve their functional capacity, quality of life, and the control of cardiovascular risk factors, more than walking because they can not achieve the ideal exercise intensity for maximal benefits by walking. This study has been designed to investigate if CHD patients get more health benefits with the supervised exercise program at the health center than with the unsupervised walking program.

DETAILED DESCRIPTION:
In order to obtain the maximal health benefits, CHD patients have to attain an exercise intensity between 60 and 85% of the maximal or symptom-limited heart rate (HR). This is not currently attained by the patients who are prescribed an unsupervised walking program.

The OBJECTIVE of this randomized clinical trial is to investigate if CHD patients improve their functional capacity and quality of life more, and control their cardiovascular risk factors better, by coming to their health centers to pedal during 30 minutes on an stationary bicycle , 3 or more times a week, with a HR monitor which makes sure that they attain HRs within the prescribed interval, and supervised by health personal, than by walking without supervision. For that purpose, low risk CHD patients from 11 Spanish health centers will be randomly assigned to a supervised exercise group (ESCAP) or to another unsupervised walking group (control). Both groups will be also provided with health education and the corresponding treatment for cardiovascular risk factor control and complication prevention by their family physicians. The average changes observed in the two groups will be compared, on the basis of intention to treat through analysis of covariance. We will use mixed-effect models to take into account intra-patients and intra-center correlation.

ELIGIBILITY:
Inclusion Criteria:

* Coronary heart disease low risk patients
* Under 80 years old

Exclusion Criteria:

* 80 years of age and over
* Patients included in cardiac rehabilitation programs
* Moderate and high risk patients
* Patients with handicaps for exercising
* Patients unable to attend the supervised exercise sessions
* Unstable angina
* Uncontrolled atrial ventricular arrhythmias
* Third degree AV block (without pacemaker)
* Uncompensated congestive heart failure
* Severe aortic stenosis
* Suspected or known dissecting aneurysm
* Active myocarditis or pericarditis
* Thrombophlebitis
* Recent embolism
* Acute systemic illness or fever
* Significant emotional distress (psychosis)
* Orthostatic blood pressure drop of >20 mm Hg with symptoms
* Uncontrolled sinus tachycardia
* Resting ST segment displacement (>2 mm)
* Uncontrolled diabetes (resting blood glucose >400 mg/dl)
* Other metabolic problems such as acute thyroiditis, hypo or hyperkalemia, hypovolemia, etc.
* Resting SBP>200 mm Hg or resting DBP>110 mm Hg

Ages: 20 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2005-01; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Functional capacity (exercise treadmill test) | 6 months follow-up

SECONDARY OUTCOMES:
Health Related Quality of life (SF-36) | 6 months follow-up
Cardiovascular risk factor control | 6 months follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Ricardo Ortega, Dr., Principal Investigator — Santa Barbara primary care center (Castilla La Mancha Health Service)
Locations (2):
- Spain (2):
  - Primary Care Research Unit of Bizkaia (Basque Health Service), Bilbao, Bizkaia
  - Santa Barbara primary care center (Castilla La Mancha Health Service), Toledo, Toledo

REFERENCES:
- [Background] Ortega Sanchez-Pinilla R. [Differences in intensity of effort between supervised and non-supervised exercise of patients with ischaemic cardiopathy]. Aten Primaria. 2004 Sep 30;34(5):265-6. doi: 10.1016/s0212-6567(04)70847-1. No abstract available. Spanish. PMID 15456577
- [Derived] Ortega R, Garcia-Ortiz L, Torcal J, Echevarria P, Vargas-Machuca C, Gomez A, Salcedo F, Lekuona I, Montoya I, Grandes G; ESCAP Group. Supervised exercise for acute coronary patients in primary care: a randomized clinical trial. Fam Pract. 2014 Feb;31(1):20-9. doi: 10.1093/fampra/cmt059. Epub 2013 Oct 19. PMID 24142481